CLINICAL TRIAL: NCT06139705
Title: Weather Sensitivity Profile and the Effects of Walking in Nature on Psychophysiological Stress Response in Individuals With Coronary Artery Disease
Brief Title: Weather Sensitivity and the Effects of Walking in Nature on Stress Response of Individuals With Coronary Artery Disease
Acronym: SENSE_NATURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Dalia Martinaitiene, Principal Investigator, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BE-2-9; S-MIP-23-114 (Other Grant/Funding Number: Research Council of Lithuania)
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease; Cardiac Rehabilitation; Nature, Human; Stress Reaction; Cognitive Function 1, Social
Keywords: coronary artery diseases; weather sensitivity; cardiac rehabilitation; nature; stress reaction; walking
MeSH Terms: conditions — Coronary Artery Disease; Fractures, Stress

STUDY DESIGN:
Intervention Model Description: After baseline measurements, the patients will be randomly assigned to either walking outdoors (OUT) or walking indoors (IN) groups. OUT group will walk in the parke. IN group will walk in a gym on a treadmill. During both interventions, the patient will be supervised by researchers. The order and sequence of measurements within each trial will be the same.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking outdoors group (OUT group) (Experimental): The OUT group will walk in natural environment.
  Interventions: Other: Walking outdoor
- Walking indoors group (IN group) (Experimental): The IN group will walk indoors.
  Interventions: Other: Walking indoor

INTERVENTIONS:
Other: Walking outdoor — The individuals will walk in park along a pre-designated route 20 min.
  Arms: Walking outdoors group (OUT group)
Other: Walking indoor — The individuals will walk in a gym on a treadmill 20 min.
  Arms: Walking indoors group (IN group)

SUMMARY:
The goal of this clinical trial is to investigate how walking in different environments affects the psychophysiological responses to the stress of individuals with coronary artery disease (CAD) according to their weather sensitivity. Awareness about the potential influence of weather sensitivity on the psychophysiological reactions to stress in patients with CAD disease may contribute to the planning and implementation of actions leading to improved medical care services and preventative measures that help to avoid the worsening of health and well-being in the future.

DETAILED DESCRIPTION:
The environment might influence one's course of a disease and health prospective through direct exposure to physical, chemical, social, and psychosocial risk factors, as well as indirectly, through behavior-related changes response to those factors. Classical risk factors only partially account for variations in the occurrence, incidence, and mortality of cardiovascular disease (CVD). Therefore, other, less-explored factors need to be taken in consideration when referring to CVD epidemiology.

The main goal of this clinical trial is to investigate how walking in different environments affects the psychophysiological responses to the stress of individuals with coronary artery disease (CAD) during rehabilitation. An experimental study will be carried out including individuals with CAD attending cardiac rehabilitation. The hypothesis is that psychophysiological reactions to stress in weather-sensitive (WS) individuals with CAD will differ from non-WS individuals when walking outdoors (in a natural environment).

To achieve the main goal, the following specific tasks will be implemented:

1. To determine how walking in a natural environment affects the psychophysiological reactions to stress in individuals with CAD.
2. To determine how walking in the gym affects the psychophysiological reactions to stress in individuals with CAD.
3. To analyse the associations between the psychophysiological reactions to stress of individuals with CAD and the walking environment, considering the sensitivity to the weather.
4. To determine the connections between mental flexibility and weather sensitivity.

The participants will be randomly assigned to either walking outdoors (OUT) or walking indoors (IN) groups. OUT group will walk in natural environment (in the park) along a pre-designated route. IN group will walk in a gym on a treadmill. The order and sequence of measurements within each trial will be the same. During both interventions, the participants will be supervised by investigators.

The idea is to increase knowledge about the impact of the natural environment on well-being and health and to provide more information to health professionals and the public. Awareness about the potential influence of weather sensitivity on the psychophysiological reactions to stress in patients with CAD disease may contribute to the planning and implementation of actions leading to improved medical care services and preventative measures that help to avoid the worsening of health and well-being in the future. Protective measures should be directed towards susceptible groups rather than the population. The outcomes of this experiment may have direct clinical applications for the use of different types of environments in cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. from 18 years and older,
2. diagnosis of CAD,
3. participation in the cardiac rehabilitation program,
4. able to hear, speak and read in Lithuanian, and
5. signed informed consent.

Exclusion Criteria:

1. coronary artery bypass graft surgery, other cardiac surgery graft,
2. cognitive or communicative disabilities or other severe comorbidities,
3. unstable cardiovascular status,
4. did not speak Lithuanian fluently,
5. did not consent in participating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Psychophysiological respond to stress | Two days
  The primary outcome is psychophysiological reaction to stress. Psychophysiological stress responses will be assessed by hemodynamic parameters and cortisol level. concentration in saliva. Hemodynamic parameters will be measured using a long-term blood pressure device, which simultaneously, continuously, and non-reactively records blood pressure, ECG, and oxygen saturation, allowing comparative analysis of several vital parameters. A long-term BP monitor will be placed on the participant in the morning, duration of measurement up to 24 hours. Cortisol levels will be measured from saliva. Saliva samples will be obtained from participants using saliva sampling tubes. Samples will then be stored at -70 zero of Celsius and cortisol levels will be determined in a licensed laboratory using commercial reagent kits. Saliva samples will be taken five times: two times a day before experiment, three times - during experiment. One sampling procedure duration up to 2 min.

SECONDARY OUTCOMES:
Weather sensitivity | up to 5 minutes
  To assess weather sensitivity, individuals will be filled in Palanga self-assessment diary for weather sensitivity (PSAD-WS). PSAD-WS is an 11-item (general) three-factor tool for collecting information regarding weather sensitivity in patients with CAD. The three subscales reflected 1) psychological symptoms, 2) cardiac symptoms and 3) physical. Also, individuals will be asked a single question: "Do you feel the weather changes?" with possible answers of "NO" or "YES".
Mental flexibility | up to 60 minutes
  Mental flexibility will be evaluated using Cambridge Neuropsychological Test Automated Battery (CANTAB). CANTAB evaluate alterations in executive function. Specifically, the following tests is used: Motor screening Task - sensorimotor function; Cambridge Gambling Test - decision making (impulsivity, risk taking); Delayed Matching to Sample - short-term visual recognition memory; Intra-Extra Dimensional Set Shift - set-shifting, mental flexibility; Match to Sample Visual Search - attention and visual searching; One Touch Stockings - spatial planning and the working memory; Rapid Visual Information Processing - sustained attention; Spatial Working Memory - working memory.

CONTACTS AND LOCATIONS:
Overall Officials: Nijole Kazukauskiene, Dr., Principal Investigator — Lithuanians Uiversity of Health Sciences
Locations (1):
- Laboratory of Behavioral Medicine, Neuroscience Institute, Lithuanian University of Health Sciences, Palanga, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gecaite J, Burkauskas J, Brozaitiene J, Mickuviene N. Cardiovascular Reactivity to Acute Mental Stress: THE IMPORTANCE OF TYPE D PERSONALITY, TRAIT ANXIETY, AND DEPRESSION SYMPTOMS IN PATIENTS AFTER ACUTE CORONARY SYNDROMES. J Cardiopulm Rehabil Prev. 2019 Nov;39(6):E12-E18. doi: 10.1097/HCR.0000000000000457. PMID 31688512
- [Background] Abrignani MG, Lombardo A, Braschi A, Renda N, Abrignani V. Climatic influences on cardiovascular diseases. World J Cardiol. 2022 Mar 26;14(3):152-169. doi: 10.4330/wjc.v14.i3.152. PMID 35432772
- [Derived] Martinaitiene D, Sampaio F, Demetrovics Z, Gjoneska B, Portacenko J, Damuleviciute A, Garbenyte-Apolinskiene T, Burkauskas J, Kazukauskiene N. A randomised controlled trial assessing the effects of weather sensitivity profile and walking in nature on the psychophysiological response to stress in individuals with coronary artery disease. A study protocol. BMC Psychol. 2024 Feb 19;12(1):82. doi: 10.1186/s40359-024-01574-3. PMID 38374158